CLINICAL TRIAL: NCT06360653
Title: a SIngle Center Study of Post-operative STEReotactic RAdiotherapY for Endometrial Cancer (SISTER-RAY)
Brief Title: a SIngle Center Study of Post-operative STEReotactic RAdiotherapY for Endometrial Cancer
Acronym: SISTER-RAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ARNAS Civico Di Cristina Benfratelli Hospital (Other)
Collaborators: Accuray Incorporated (Industry)
Responsible Party: Principal Investigator, Francesco Cuccia, MD, Principal Investigator, ARNAS Civico Di Cristina Benfratelli Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 76CIVICO2023
Record Dates: First submitted 2024-04-05; First posted 2024-04-11 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; radiotherapy; sbrt
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients with endometrial cancer (stage IB-IIIC1) with histological and molecular features that require adjuvant external beam radiotherapy alone or in combination with chemotherapy and/or brachytherapy. Adjuvant radiotherapy will be performed with stereotactic body radiotherapy schedule of 30 Gy in 5 sessions.
  Interventions: Radiation: Stereotactic Post-operative Radiotherapy for Endometrial Cancer

INTERVENTIONS:
Radiation: Stereotactic Post-operative Radiotherapy for Endometrial Cancer — Patients candidate to receive adjuvant radiotherapy will be assigned to a shorter schedule of 30 Gy in 5 sessions.

SUMMARY:
The primary endpoint of the present prospective study is to assess the outcomes in terms of acute toxicity of post-operative stereotactic radiotherapy for endometrial cancer

DETAILED DESCRIPTION:
Endometrial cancer represents the sixth global female cancer, and adjuvant radiotherapy has a main role in the management of these patients.

This treatment usually covers the surgical bed, the upper portion of the vagina and the pelvic lymph nodes. In the last decades, the technological progress has allowed clinicians to offer a more accurate planning and delivery of the treatment with modern IMRT-IGRT techniques.

Nonetheless, radiotherapy regimens were still based on 25-30 fractions schedules. More recently, similarly to other oncological settings like prostate, breast or rectal cancer, 5-fractions schedules have been considered as potentially useful also in this setting.

On this purpose, this study aims to investigate the feasibility of a shorter adjuvant radiotherapy treatment for endometrial cancer, by assessing acute and late toxicity, quality of life and clinical outcomes.

ELIGIBILITY:
* Age 18-80 years
* ECOG PS ≤ 2 or KPS ≥ 70%
* Patients diagnosed with endometrial cancer (endometrioid, serous cell, clear cell, carcinosarcoma) FIGO stage IB-IIIC1 candidate to post-operative external beam radiotherapy, based on molecular and histological findings
* Indications for chemotherapy and/or brachytherapy are not exclusion criteria for the purpose of the study
* Written Informed Consent

Exclusion Criteria:

* Prior pelvic radiotherapy
* Para-aortic lymph nodes involvement
* ECOG PS ≥ 3
* Any diagnosis of inflammatory bowel disease (both active or quiescent)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Acute G3 or higher Gastrointestinal and Genitourinary Toxicity | From the end of treatment to a time interval of 12 weeks
  The number of any G3 or higher adverse event occurring within 90 days from the end of radiotherapy and assessed according to the CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Late Gastrointestinal and Genitourinary Toxicity | From enrollment to a follow-up time of 5 years
  The number of any G3 or higher adverse event occurring after 90 days from the end of radiotherapy and assessed according to the CTCAE v5.0 criteria
Distant Progression Free Survival | From enrollment to a follow-up time of 5 years
  The rate of distant failure of the disease in all the participants enrolled for adjuvant SBRT
Local Control | From enrollment to a follow-up time of 5 years
  The rate of local failure of the disease in all the participants enrolled for adjuvant SBRT
Overall Survival | From enrollment to a follow-up time of 5 years
  The rate of death events in the cohort of patients enrolled
Overall Quality of Life | From enrollment to a follow-up time of 5 years
  The mean values of Quality of life questionnaires performed at baseline and at 3-6-12-18-24-36- 48-60 months from the end of treatment, with the QLQ-C30 and QLQ-EN24 fulfilled by all patients enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- ARNAS Civico Hospital, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung E, Gladwish AP, Davidson M, Taggar A, Velker V, Barnes E, Mendez L, Donovan E, Gien LT, Covens A, Vicus D, Kupets R, MacKay H, Han K, Cheung P, Zhang L, Loblaw A, D'Souza DP. Quality-of-Life Outcomes and Toxic Effects Among Patients With Cancers of the Uterus Treated With Stereotactic Pelvic Adjuvant Radiation Therapy: The SPARTACUS Phase 1/2 Nonrandomized Controlled Trial. JAMA Oncol. 2022 Jun 1;8(6):1-9. doi: 10.1001/jamaoncol.2022.0362. PMID 35420695
- [Background] Musunuru HB, D'Alimonte L, Davidson M, Ho L, Cheung P, Vesprini D, Liu S, Chu W, Chung H, Ravi A, Deabreu A, Zhang L, Commisso K, Loblaw A. Phase 1-2 Study of Stereotactic Ablative Radiotherapy Including Regional Lymph Node Irradiation in Patients With High-Risk Prostate Cancer (SATURN): Early Toxicity and Quality of Life. Int J Radiat Oncol Biol Phys. 2018 Dec 1;102(5):1438-1447. doi: 10.1016/j.ijrobp.2018.07.2005. Epub 2018 Jul 31. PMID 30071295
- [Background] Klopp AH, Moughan J, Portelance L, Miller BE, Salehpour MR, Hildebrandt E, Nuanjing J, D'Souza D, Souhami L, Small W Jr, Gaur R, Jhingran A. Hematologic toxicity in RTOG 0418: a phase 2 study of postoperative IMRT for gynecologic cancer. Int J Radiat Oncol Biol Phys. 2013 May 1;86(1):83-90. doi: 10.1016/j.ijrobp.2013.01.017. PMID 23582248